CLINICAL TRIAL: NCT00833274
Title: Evaluation of Apathy Using Attentional Reaction Test in Neurodegenerative Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-CIR-01
Record Dates: First submitted 2009-01-28; First posted 2009-02-02 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Using a computerized test, each patient is asked to press a button (mouse of the computer) each time the screen of the computer becomes completely white.
  Interventions: Behavioral: computerized test

INTERVENTIONS:
Behavioral: computerized test — Using a computerized test, each patient is asked to press a button (mouse of the computer) each time the screen of the computer becomes completely white.

SUMMARY:
Apathy, defined as a lack of motivation in behaviour, cognition and affect, is common in neurodegenerative diseases. Specific scales are available for the evaluation of apathy but it lacks objective evaluation methods.

The aim of this study is to evaluate the changes in reaction time task according to the presence or absence of reward stimulation and to assess the relation between these performances and apathy scales.

DETAILED DESCRIPTION:
MATERIAL: 13 patients with Mild Cognitive Impairment (MCI), 15 patients with Alzheimer's disease (AD) and 91 elderly healthy subjects were enrolled. A computerized test using the experiment software E-prime® was designed to assess reaction times (in ms) in different experimental conditions after a training trial (neutral, stimulation, stress, stimulation after stress, extinction) and relation between the performances to the test and the Apathy Inventory (AI) scores (lack of initiative, lack of interest, emotional blunting) were observed.

METHOD: Using a computerized test, each patient is asked to press a button (mouse of the computer) each time the screen of the computer becomes completely white. After pressing the button, a randomized colorized geometric figure appears on the screen, and disappears automatically after a few seconds, replaced by a new white screen. Reaction time (in ms) between a white screen and a press of the button is analysed. After a training trial, reaction times are analysed in different experimental conditions: neutral - stimulation1 (patient gets points when pressing the button) - stress (alarm) - stimulation2 (patient gets points when pressing, after the stress trial) - extinction (similar to neutral condition).

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients with diagnosis of Alzheimer's Disease according to DSM-IV criteria
* MMSE >20

Exclusion Criteria:

* None
* Motor or psychiatric disorders

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Reaction times (ms), using a computerized test | one time point, at day 0 (day of inclusion) during the computerized test

SECONDARY OUTCOMES:
Apathy severity, using a specific apathy scale (Apathy Inventory) | one time point, at day 0 (day of inclusion), during the visit

CONTACTS AND LOCATIONS:
Locations (1):
- CM2R, Nice University Hospital, Nice, France